CLINICAL TRIAL: NCT02403089
Title: Ontogeny of MAIT Cells in Neonates and Hematopoietic Stem Cell Transplant Recipients
Acronym: NEOMAIT
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: NI14006
Record Dates: First submitted 2015-03-06; First posted 2015-03-31 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2018-02

CONDITIONS: Term and Preterm Neonates (24-41 Weeks Gestational Age); Hematopoietic Stem Cell Transplant Recipient Children
Keywords: MAIT (Mucosal-Associated Invariant T) cells; Gut microbiota; Preterm birth; Hematopoietic stem cell transplantation; Microbial infections
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — funds tubes samples taken as part of routine care for newborns and in allograft recipients children will be recovered. Mononuclear cells from cord blood will be isolated and stored in liquid nitrogen in the laboratory of Immunology before achieving functional tests.
  • Rectal swabs and gastric aspirates aliquots made as part of routine care for newborns, and rectal swabs made as part of routine care in HSCT allograft recipients, will be stored at -80 ° C in the laboratory of Immunology.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- neonates: neonates 24-41 weeks gestational age
  Interventions: Other: Tubes fund recovery blood count
- children: hematopoietic stem cell transplant recipient children (< 18 years old, donor source: cord blood or genoidentical donor)
  Interventions: Other: the rest of the blood test and stool sample

INTERVENTIONS:
Other: Tubes fund recovery blood count — Tubes fund recovery of blood counts among newborns
  Groups: neonates
Other: the rest of the blood test and stool sample — blood samples on the recovery kinetics after transplant. The rest of the blood test and stool sample done as part of a routine examination.
  Groups: children

SUMMARY:
The objective of this study is 1/ to determine the rate and kinetics of MAIT cell expansion and maturation in neonates in relation with gestational age, and in HSCT recipient children in relation with the source of donor stem cells, 2/ to correlate gut microbiota diversity and function with MAIT cell maturation and function in neonates and HSCT recipients; and 3/ to link MAIT cells and gut microbiota composition with microbial infections and severe intestinal inflammatory events in term and preterm neonates, and in HSCT recipients

DETAILED DESCRIPTION:
The mucosa-associated invariant T (MAIT) cells are innate-like T cells with restricted T cell receptor (TCR) usage, which are preferentially localized in mucosal tissues and respond to microbial infection by rapidly producing cytokines and cytotoxic effectors. They recognize the non-classical related molecule (MR1). MAIT cells react against a newly identified class of antigens presented by MR1: Riboflavin (Rib) precursors, which are found in most bacteria and yeasts. Currently, very little is known about the ontogeny of MAIT cells in the human, because of the difficulty to follow longitudinally their development. Cross-sectional studies have identified only the initial (cord blood) and final (adult subjects) steps of human MAIT cell maturation program. Moreover, there are no data on relationships between human MAIT cell expansion and maturation, and gut microbiota development. Given the potential importance of MAIT cells in protection from microbial infections at epithelial surfaces, we will investigate the maturation dynamics of MAIT cells in relation with gut microbiota diversity and function in two clinical settings characterized by a high predisposition to severe microbial infections before the establishment of protective adaptive immunity, namely i/ the neonatal period and ii/ the early immune reconstitution period following allogeneic hematopoietic stem cell transplantation (HSCT) in children. Our study will combine multiparametric phenotypic and functional characterization of MAIT cells with the use of new molecular microbiota analytic methodology (high throughput sequencing, metagenomics, Rib microbiology) to determine how the presence or functionality of MAIT cells is influenced by the gut microbiota.

Our consortium is composed of three independent research teams, experts in innate immunity, microbial ecology and MAIT cell biology, three independent clinical teams providing exceptional resources to patient samples, and one team providing expertise for methodology and statistical analysis. Their synergistic interaction will offer the various complementary expertise that is necessary for this project.

This project will decipher how MAIT cell numbers or functions are influenced by the gut microbiota composition, and reciprocally, how MAIT cells regulate or control expansion of gut microbiota components competing with opportunistic or pathogenic bacteria or responsible for infections. Ultimately, this study will determine how and when gut microbiota and MAIT cell interactions are involved in the control of severe infectious or intestinal inflammatory events in high risk infants, an indispensable step to design predictive biomarkers and ultimately propose new therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* neonates 24-41 weeks gestational age
* hematopoietic stem cell transplant recipient children (< 18 years old, donor source: cord blood or genoidentical donor)

Exclusion Criteria:

* neonates : chromosomal abnormalities detected before birth
* source of HSCT: phenol-identical donors

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: newborns hospitalized in the Neonatal Intensive Care Unit of the Hospital Robert Debré and grafted children hospitalized in the Hematology-Immunology Pediatric Service of the Hospital Robert Debré
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
MAIT cell numbering neonates after birth | to 60days
  Absolute number, percentage and phenotype of MAIT cells by flow cytometry in the circulating blood after birth according to gestational age and / or maternal-fetal infections (IMF), or after allogeneic HSCT according to the origin of HSCs.

SECONDARY OUTCOMES:
Absolute number of MAIT | to 60days
  Absolute number and percentage of MAIT among mothers of infants on the day of delivery and in geno-identical donors before transplantation.
Absolute number of other immune cell populations | to 60 days
  Absolute number and percentage of other immune cell populations by flow cytometry on the same blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Biran Valérie, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France

REFERENCES:
- [Result] Ben Youssef G, Tourret M, Salou M, Ghazarian L, Houdouin V, Mondot S, Mburu Y, Lambert M, Azarnoush S, Diana JS, Virlouvet AL, Peuchmaur M, Schmitz T, Dalle JH, Lantz O, Biran V, Caillat-Zucman S. Ontogeny of human mucosal-associated invariant T cells and related T cell subsets. J Exp Med. 2018 Feb 5;215(2):459-479. doi: 10.1084/jem.20171739. Epub 2018 Jan 16. PMID 29339446
- [Derived] Tourret M, Talvard-Balland N, Lambert M, Ben Youssef G, Chevalier MF, Bohineust A, Yvorra T, Morin F, Azarnoush S, Lantz O, Dalle JH, Caillat-Zucman S. Human MAIT cells are devoid of alloreactive potential: prompting their use as universal cells for adoptive immune therapy. J Immunother Cancer. 2021 Oct;9(10):e003123. doi: 10.1136/jitc-2021-003123. PMID 34615705